CLINICAL TRIAL: NCT05886660
Title: Optimizing the Combination of Intranasal Scopolamine and Sensory Augmentation to Mitigate G-transition Induced Motion Sickness and Enhance Sensorimotor Performance
Brief Title: Combination of Intranasal Scopolamine and Sensory Augmentation to Mitigate G-transition Induced Motion Sickness and Enhance Sensorimotor Performance
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Repurposed Therapeutics, Inc. (Industry)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NASA 0354 (Aim 1)
Record Dates: First submitted 2023-04-17; First posted 2023-06-02 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Motion Sickness, Space; Motion Sickness; Sea Sickness
Keywords: wave motion; eye-hand coordination; artificial horizon
MeSH Terms: conditions — Space Motion Sickness; Motion Sickness | interventions — Scopolamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: A randomized double-blind (subjects and test operators) cross-over design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DPI-386 Nasal Gel (Experimental): DPI-386 Nasal Gel, 0.4 mg
  Interventions: Drug: DPI-386 Nasal Gel
- Placebo Comparator (Experimental): Placebo Nasal Gel
  Interventions: Drug: Placebo Nasal Gel
- DPI-386 Nasal Gel and Sensory Augmentation DPI-386 Nasal Gel, 0.4 mg (Experimental): 8-Channel K-Tactile Belt, Engineering Acoustics, Inc., Casselberry, FL
  Interventions: Drug: DPI-386 Nasal Gel
- Placebo Comparator and Sensory Augmentation Placebo Nasal Gel (Experimental): 8-Channel K-Tactile Belt, Engineering Acoustics, Inc., Casselberry, FL
  Interventions: Drug: Placebo Nasal Gel

INTERVENTIONS:
Drug: DPI-386 Nasal Gel — Subjects will self-administer DPI-386 Nasal Gel.
  Other Names: scopolamine
  Arms: DPI-386 Nasal Gel
Drug: Placebo Nasal Gel — Subjects will self-administer Placebo Nasal Gel.
  Arms: Placebo Comparator
Drug: DPI-386 Nasal Gel — Subjects will self-administer DPI-386 Nasal Gel. Vibrotactile feedback of tilt direction and magnitude will be provided on a sensory augmentation belt worn by the subject.
  Other Names: scopolamine
  Arms: DPI-386 Nasal Gel and Sensory Augmentation DPI-386 Nasal Gel, 0.4 mg
Drug: Placebo Nasal Gel — Subjects will self-administer Placebo Nasal Gel.
  Vibrotactile feedback of tilt direction and magnitude will be provided on a sensory augmentation belt worn by the subject.
  Arms: Placebo Comparator and Sensory Augmentation Placebo Nasal Gel

SUMMARY:
The primary specific aim is to evaluate the use of intranasal scopolamine gel and sensory augmentation as an integrated countermeasure to mitigate motion sickness and enhance sensorimotor performance. The proposed intranasal scopolamine gel formulation (Defender Pharmaceuticals, Inc.) offers a safe non-invasive method to self-administer with a rapid onset of action. This study involves a comparison of motion sickness outcome measures when administering intranasal scopolamine gel versus placebo (Aim 1a), and then when administering intranasal scopolamine gel versus placebo with a sensory augmentation belt (Aim 1b).

DETAILED DESCRIPTION:
The primary specific aim is to evaluate the use of intranasal scopolamine gel (DPI-386) and sensory augmentation (SA) as an integrated countermeasure to mitigate motion sickness and enhance sensorimotor performance. The proposed intranasal scopolamine gel formulation (Defender Pharmaceuticals, Inc.) offers a safe non-invasive method to self-administer with a rapid onset of action. The proposed sensory augmentation will utilize vibrotactile feedback of pitch and roll tilt using a portable belt (Engineering Acoustics, Inc.). The investigators will utilize exposure to simulated capsule wave motion on a 6DOF platform to provide an operationally relevant platform to induce motion sickness and impair performance on functional tasks. The investigators hypothesize that the combination of intranasal scopolamine gel and sensory augmentation of Earth vertical will be more effective to mitigate motion sickness and improve task performance than when administered separately. Using a randomized double-blind cross-over design, the investigators will compare motion sickness symptom severity and time to endpoint (symptom level defined as severe malaise) in 30 subjects during exposure to simulated wave motion on a 6DOF platform inside of a crew capsule mockup. The investigators will compare four conditions: (1) intranasal scopolamine gel (0.4 mg) with sensory augmentation, (2) intranasal scopolamine gel (0.4 mg) without sensory augmentation, (3) placebo control with sensory augmentation, and (4) placebo control without sensory augmentation. The wave motion stressor will begin 30 min post drug administration and will not exceed 45 min in duration. Performance on a series of functional tasks (dual-task tracking and eye-hand target acquisition) will be performed pre, during, immediately post, and following 15 min of recovery of each test. The bioavailability of scopolamine for each session will be estimated from plasma concentrations obtained at drug administration and then every 15 min up to 2-hr post-dosage. Subjective side effects and performance on the Psychomotor Vigilance Test (PVT) will also be obtained at 15 min intervals.

A small pilot study including 10 subjects tested once each will be performed to verify the experimental protocol including that the simulated capsule wave motion will provoke motion sickness symptoms. These pilot sessions will not include the medication nor the blood sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should be minimally susceptible to provocative motion as evidenced by at least two responses on the Motion Sickness Susceptibility Questionnaire of "Sometimes" or "Frequently."
2. No participants should have neurologic, vestibular or autonomic disorders, or medical conditions that could be worsened by scopolamine (narrow-angle glaucoma or urinary retention
3. Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) negative test, confirmed by Food and Drug Administration (FDA) authorized COVID-19 test < 7 days prior to study drug administration or no COVID 19 symptoms up to 10 days prior to study drug administration.

Exclusion Criteria:

1. Subjects will be excluded if they are taking other drugs that are capable of causing CNS effects such as antihistamines, tricyclic antidepressants, and muscle relaxants or have hypersensitivity to scopolamine or other belladonna alkaloids or to any ingredient or component in the formulation or delivery system.
2. Pregnant women are excluded from participation. Women of child-bearing potential will be offered a pregnancy screening test and excluded with a positive test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Motion sickness (MS) symptom severity using Pensacola Diagnostic Index (PDI) scale | 45 minutes
  The PDI scale ranges from 0 to 16 with higher numbers reflecting greater symptom severity (in this study a PDI score of 8 will be used as a motion sickness (MS) endpoint).
  During each session, the primary motion sickness symptoms will be recorded every minute during the capsule wave motion stimulation through the MS endpoint (PDI score ≥ 8 points) up to 45 min total.

SECONDARY OUTCOMES:
Motion sickness symptom severity using a Subjective Discomfort Rating (SDR) | 45 minutes
  The SDR scale ranges from 0-20 with higher numbers reflecting greater symptom severity (20 = vomiting). This will be recorded at the same interval as the PDI score.
Time to MS endpoint (based on PDI score of 8 points) | 45 minutes
  The time to MS endpoint will be recorded once per session, range of 0-45 with higher numbers reflecting less motion sickness susceptibility.
Performance measures: response time | 45 minutes
  Response time during eye-hand coordination tasks will be recorded once every 15 min of stimulation (up to three measures per session) with the shorter response representing better performance.
Performance measures: error | 45 minutes
  Response error during eye -hand coordination tasks will be recorded once every 15 min of stimulation (up to three measures per session), with lower error representing better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Scott J Wood, PhD, Principal Investigator — National Aeronautics and Space Administration (NASA)
Locations (1):
- NASA Johnson Space Center Neuroscience Laboratory, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No